CLINICAL TRIAL: NCT06466187
Title: A Phase 1 Open-label, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of SGN-MesoC2 in Subjects With Advanced Solid Tumors
Brief Title: A Study of SGN-MesoC2 in Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C5991001; SGNMesoC2-001 (Other: Alias Study Number)
Record Dates: First submitted 2024-06-11; First posted 2024-06-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Pancreatic Adenocarcinoma; Colorectal Neoplasms; Mesothelioma; Other Solid Tumors; Endometrial
Keywords: NSCL; Lung Neoplasm; Cancer of Ovary; Ovarian Cancer; Colorectal Cancer; Colorectal Tumors; Endometrial; Seattle Genetics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Colorectal Neoplasms; Mesothelioma; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-08052666 (Experimental): PF-08052666 monotherapy
  Interventions: Drug: PF-08052666

INTERVENTIONS:
Drug: PF-08052666 — Given into the vein (IV; intravenously)
  Other Names: HBM9033; SGN-MesoC2

SUMMARY:
This clinical trial is studying advanced solid tumors. Solid tumors are cancers that start in a part of your body like your lungs or liver instead of your blood. Once tumors have grown bigger in one place but haven't spread, they're called locally advanced. If your cancer has spread to other parts of your body, it's called metastatic. When a cancer has gotten so big it can't easily be removed or has spread to other parts of the body, it is called unresectable. These types of cancer are harder to treat.

Patients in this study must have cancer that has come back or did not get better with treatment. Patients must have a solid tumor cancer that can't be treated with standard of care drugs.

This clinical trial uses an experimental drug called PF-08052666/SGN-MesoC2. PF-08052666/SGN-MesoC2 is a type of antibody-drug conjugate (ADC). ADCs are designed to stick to cancer cells and kill them. They may also stick to some normal cells.

This study will have 3 parts. Part A and Part B of the study will find out how much PF-08052666/SGN-MesoC2 should be given to participants. Part C will use the information from Parts A and B to see if PF-08052666/SGN-MesoC2 is safe and if it works to treat solid tumor cancers.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Histologically- or cytologically-confirmed metastatic or locally advanced unresectable platinum-resistant ovarian cancer, NSCLC, pancreatic ductal adenocarcinoma, endometrial cancer, colorectal cancer, or mesothelioma, who have relapsed or progressed following standard therapies, or for which no standard therapies are available.
* An Eastern Cooperative Oncology Group performance status score of 0 or 1.
* At least 1 measurable lesion at baseline based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1).
* Archival tumor tissue or a fresh tumor biopsy during the screening period.
* Adequate hepatic, renal and bone marrow function.
* Participants must not have received more than 2 lines of cytotoxic systemic therapy in the metastatic setting (Parts B and C only).

Exclusion Criteria:

* Previously received or currently receiving any systemic anticancer therapy or focal radiotherapy within 4 weeks prior to the first dose of MesoC2 or within 2 weeks prior to the first dose of MesoC2 if the underlying disease had progressed on treatment.
* Prior anti-MSLN antibody or MSLN-directed ADC (Part C only).
* Unresolved toxicities from prior therapy greater than NCI CTCAE v5.0 grade 1 at the time of study treatment (except alopecia).
* Inadequate hepatic dysfunction, renal function, or hematologic abnormalities.
* Previously untreated brain metastases. Participants who received radiation or surgery for brain metastases are eligible if therapy was completed at least 4 weeks prior to study treatment initiation, and there was no evidence of central nervous system progression nor requirements for chronic corticosteroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Through 30-37 days after the last dose of study treatment, 48 Months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants with laboratory abnormalities | Through 30-37 days after the last dose of study treatment, 48 Months
Number of participants with dose modifications | Up to 4 months
  Frequency of dose modifications (eg, dose delay, treatment interruptions, dose reductions and treatment discontinuations) due to AEs
Number of participants with dose-limiting toxicities (DLTs) | Cycle 1 (21 days)
  Incidence of dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Objective response rate (ORR) | Approximately 1 year 4 months
  ORR is defined as the proportion of participants in the relevant analysis set with best response of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Best response | Approximately 1 year 4 months
  The best timepoint response achieved for the subject during the protocol specified period according to RECIST V1.1.
Duration of response (DOR) | Approximately 1 year 4 months
  DOR is defined as the time interval from first occurrence of documented objective response to the time of progressive disease (PD) according to RECIST v1.1 or death from any cause, whichever comes first.
Disease control rate (DCR) | Approximately 1 year 4 months
  DCR is defined as the proportion of participants with best response of CR, PR or stable disease (SD) according to RECIST v1.1.
Progression-free survival (PFS) | Approximately 1 year 4 months
  PFS is defined as the time from first dosing to the first occurrence of PD according to RECIST v1.1 or death from any cause, whichever comes first.
Overall survival (OS) | Approximately 1 year 4 months
  Overall survival (OS) defined as the time from first dosing to death.
Pharmacokinetic (PK) parameter - Area under the serum concentration (AUC) | Cycles 1, 2, and 3 (each cycle is up to 21 days)
Pharmacokinetic (PK) parameter - Maximum serum concentration (Cmax) | Cycles 1, 2, and 3 (each cycle is up to 21 days)
Pharmacokinetic (PK) parameter - Time to reach maximum serum concentration (Tmax) | Cycles 1, 2, and 3 (each cycle is up to 21 days)
Pharmacokinetic (PK) parameter - Half-life | Cycles 1, 2, and 3 (each cycle is up to 21 days)
Number of participants with antidrug antibodies | Cycles 1, 2, and 3 (each cycle is up to 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - The Board of Trustees of the University of Alabama for the University of Alabama at Birmingham, Birmingham, Alabama
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - The University of Kansas Hospital Cambridge North Tower A, Kansas City, Kansas
  - The University of Kansas Hospital, Kansas City, Kansas
  - The University of Kansas Medical Center Medical Office Building, Kansas City, Kansas
  - The University of Kansas Cancer Center - Indian Creek Campus, Overland Park, Kansas
  - The University of Kansas Cancer Center - Westwood, Westwood, Kansas
  - The University of Kansas Cancer Center, Investigational Drug Services, Westwood, Kansas
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Sarah Cannon Research Institute - Pharmacy, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - START San Antonio, LLC, San Antonio, Texas
  - START Mountain Region, LLC, Salt Lake City, Utah
  - START Mountain Region, West Valley City, Utah
- Canada (4):
  - University Health Network, Toronto, Ontario
  - University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario
  - The Research Institute of the McGill University Health Centre, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5991001